CLINICAL TRIAL: NCT03228641
Title: A Prospective, Multi-center, Randomized Pilot Study for the Safety and Efficacy of a GEN II Micro-coring Device for the Treatment of Wrinkles and Skin Laxity in the Pre-auricular Area and Mid to Lower Face
Brief Title: Evaluation of Safety and Efficacy of Micro-coring Device for Treatment of Facial Wrinkles and Skin Laxity
Acronym: AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 700-00001
Record Dates: First submitted 2017-02-14; First posted 2017-07-25 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Wrinkle; Facial and Neck Skin Laxity
Keywords: skin rejuvenation; wrinkle removal; skin laxity reduction
MeSH Terms: conditions — Facies

STUDY DESIGN:
Masking Description: subject is blinded to the needle gauge and density of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- micro-excisional skin removal (Experimental): Facial and neck wrinkles will be treated with micro-excisional skin removal
  Interventions: Device: micro-excisional skin removal with coring needle

INTERVENTIONS:
Device: micro-excisional skin removal with coring needle
  Other Names: micro-coring, micro-excisional skin removal

SUMMARY:
A pilot study is designed to evaluate safety and efficacy of the Micro-Coring (MC) technology for treatment of facial wrinkles. MC device employs hollow coring needles that enable safe, rapid, and effective full-thickness small skin cores (200-500 microns in diameter) removal initiating a skin repair process through formation of new collagen and elastin fibers (skin rejuvenation).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, single blind, bilateral paired study evaluating the safety, tolerability and preliminary effectiveness of a micro-coring device for removal of excess skin using 2 needle gauges (22G, 24G,) at densities (percent of skin removed per 1cm2) of 2.5-10% in subjects with mid- and lower- face skin laxity manifested by moderate-to-severe mid and lower cheek wrinkles, deepening of the nasolabial folds at rest; prominence of marionette lines at rest; downturn of the oral commissures at rest, sagging of the skin at the jawline at rest. Subjects are blinded to needle gauge and density.

There will be two cohorts of subjects: one group of subjects will receive a single treatment and the second - multiple treatments. All subjects will be followed for 180 days with several intermediate visits at 3, 7, 30, 60, and 90-days.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type 1, 2, or 3 as assessed by Investigator
* One or more of the following conditions assessed by Investigator using provided Severity Scales:

  * Nasolabial fold severity at rest ≥2 and ≤4;
  * Marionette line prominence at rest ≥2 and ≤4;
  * Oral commissure drooping at rest ≥2 and ≤4;
  * Jawline sagging at rest ≥2 and ≤4 .
  * Moderate-to-Severe wrinkles at rest at least in one of the following areas - the upper lip, chin and cheeks.

Exclusion Criteria:

* Lesions suspicious for any malignancy or the presence of actinic keratosis, melasma, vitiligo, cutaneous papules/nodules or active inflammatory lesions in the areas to be treated
* History of keloid formation or hypertrophic scarring
* History of trauma or surgery to the treatment areas in the past 6 months
* Scar present in the areas to be treated
* Silicone or synthetic material injections in the areas to be treated
* Injection of FDA-approved dermal fillers in the past two years
* Injection of fat in the past year
* History of treatment with dermabrasion, ablative laser, or radiofrequency in the past year
* History of treatment with non-ablative laser in the past 6 months
* History of treatment with botulinum toxin injections in the areas to be treated within the prior 6 months
* Active smokers (0.5 pack/day) or having quit within 3 months prior to treatment
* Active, chronic, or recurrent infection
* History of compromised immune system or currently being treated with immunosuppressive agents
* History of sensitivity to analgesic agents, Aquaphor®, topical or local anesthetics (e.g., lidocaine, benzocaine, procaine) or chlorhexidine, povidone-iodine or epinephrine
* Excessive sun exposure and use of tanning beds or tanning creams within 30 days prior to treatment
* Treatment with aspirin or other blood thinning agents within 14 days prior to treatment
* History or presence of any clinically significant bleeding disorder
* Co-morbid condition that in the Investigator's opinion could limit ability to participate in the study or to comply with follow-up requirements
* History of drug and/or alcohol abuse
* Any issue that, at the discretion of the Investigator, would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent
* Treatment with an investigational device or agent within 30 days before treatment or during the study period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
improvement in wrinkle appearance | 60 and 90 days
  One grade or better improvement in score on Wrinkle Severity Scale

SECONDARY OUTCOMES:
improvement in skin laxity | up to 180 days
  One grade or better improvement in score on Laxity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michail M Pankratov, MD, PhD, Study Director — Senior Vice President of Clinical & Regulatory Affairs; Patricia E Krantz, Study Director — Director of Clinical Operations
Locations (5):
- United States (5):
  - Laser & Skin Center of Northern CA, Sacramento, California
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Laser & Skin Surgery Center of NY, New York, New York
  - Nashville Center for Laser & Facial Surgery, Nashville, Tennessee
  - Dr A Jay Burns Cosmetic Surgery, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical data analysis will be summarized in the Clinical Study Report and later submitted for publication in the peer-reviewed journal

REFERENCES:
- [Result] Fernandes JR, Samayoa JC, Broelsch GF, McCormack MC, Nicholls AM, Randolph MA, Mihm MC, Austen WG Jr. Micro-mechanical fractional skin rejuvenation. Plast Reconstr Surg. 2013 Feb;131(2):216-223. doi: 10.1097/PRS.0b013e3182789afa. PMID 23357983
- [Result] Russe E, Purschke M, Farinelli WA, Wang Y, Doukas AG, Limpiangkanan W, Sakamoto FH, Tam J, Wechselberger G, Anderson RR. Micro-fractional, directional skin tightening: A porcine model. Lasers Surg Med. 2016 Mar;48(3):264-9. doi: 10.1002/lsm.22444. Epub 2015 Dec 2. PMID 26627306